CLINICAL TRIAL: NCT06838065
Title: Rehabilitation Management for Patients with Multiple Myeloma: a Retrospective Observational Study on Bone Fragility and Rehabilitation Needs in This Patient Population
Brief Title: Rehabilitation Management for Patients with Multiple Myeloma
Acronym: FKTMM2022
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 418/2022/OSS/AUSLRE
Record Dates: First submitted 2025-01-22; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma Bone Lesions; Multiple Myeloma (MM)
Keywords: multiple myeloma; skeletal-related events; rehabilitation
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with a new diagnosis of Multiple Myeloma: who were managed by the Hematology Department in 2019, 2020, and 2021

SUMMARY:
Multiple myeloma (MM) is the second most common blood cancer. Bone involvement is very common in these patients: it is estimated that between 80% and 90% will develop bone lesions during the course of the disease. This represents a potential risk of fragility and pain, significantly impacting the patient's functional status and therefore worsening their quality of life. [1] The presence of bone lesions also represents a risk for the development of Skeletal-Related Events (SREs), which can include: pathological fractures, vertebral compression that causes spinal cord compression, and the need for surgery or radiotherapy to treat the bone lesions. It is important to monitor and manage SREs as they are associated with increased mortality.

With the improvement of treatments and increased survival rates, more and more patients require rehabilitation management, which includes therapeutic education, the prescription of orthoses/aids, and specific rehabilitation programs to address fatigue or cope with major events such as SREs. Also frequently needed are guidelines regarding safe physical activity and support for returning to work or resuming satisfying social participation.

In many MM patients, bone involvement represents a challenge for the rehabilitation specialist, who must be able to perform an accurate assessment of the risks and benefits of treatment to avoid exposing the patient to unnecessary risks or complications. Managing the patient within a multidisciplinary team of specialists can improve the accuracy of the overall assessment and therapeutic recommendations. The aim of our study is to retrospectively analyze patients with a new diagnosis of MM who were managed by the Hematology Department in 2019, 2020, and 2021, in order to describe and evaluate any SREs, as well as some clinical and rehabilitation data.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is the second most common blood cancer. Bone involvement is very common in these patients: it is estimated that between 80% and 90% will develop bone lesions during the course of the disease. This represents a potential risk of fragility and pain, significantly impacting the patient's functional status and thus worsening their quality of life.

Furthermore, the presence of bone lesions represents a risk for the development of Skeletal-Related Events (SREs), which can include pathological fractures, vertebral compressions causing spinal cord compression, and the need for surgery or radiotherapy to treat bone lesions. It is important to monitor and manage SREs as they are associated with an increased risk of mortality.

With improvements in treatment and increased survival, more and more patients require rehabilitative care, which includes therapeutic education, the prescription of orthoses/aids, the implementation of specific rehabilitation programs to counter fatigue, or to address major events such as SREs. Equally important are guidelines regarding safe physical activity and support for returning to work or resuming satisfying social participation.

In many MM patients, bone involvement represents a challenge for the rehabilitation professional, who must be able to make an accurate assessment of the risks and benefits of treatment to avoid exposing the patient to inappropriate risks or complications. Caring for the patient within a multidisciplinary team of specialists can improve the accuracy of the overall assessment and therapeutic recommendations.

The aim of our study is to retrospectively analyze patients with a new diagnosis of MM who were managed by the Hematology Department in the years 2019, 2020, and 2021, in order to describe and assess any SREs, as well as some clinical and rehabilitative data.

ELIGIBILITY:
Inclusion Criteria:

* New Diagnosis of Multiple Myeloma in 2019,2020 or 2021
* Older then 18 years

Exclusion Criteria:

* Absence of even one inclusion criterion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with new Diagnosis of Multiple Myeloma in 2019,2020 or 2021 managed by the Hematology Department.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Number of patients who experienced a Skeletal-Related Event (SRE) in the first 2 years from MM diagnosis | SREs will be detected in the period including 60 days before MM diagnosis to 24 months after diagnosis
  The Presence of SREs (pathological fractures, radiation to bone, bone surgery or spinal cord compression) will be recorded from clinical databases for each patient, considering the period including 60 days before MM diagnosis to 24 months after diagnosis.
Number pf patients who underwent Hospitalization due to SREs | between 60 days before MM diagnosis and 24 months after MM diagnosis
  Record if the patient was hospitalized due to complications from SREs, considering this timeframe: between 60 days before MM diagnosis and 24 months after MM diagnosis.
Number of patients reporting a pathological fracture, number of patients who needed radiation to bone, number of patients who underwent bone surgery, number of patients with spinal cord compression. | between 60 days before MM diagnosis and 24 months after MM diagnosis
  SREs are classified it as:
  * pathological fractures
  * spinal cord compression
  * surgical stabilization of bone
  * radiotherapy on bone This outcome will record how many patients experienced each of these SREs, in different moments of MM timeline.
  We will specify if it is a:
  * baseline SREs if patients experienced it within 60 days before MM diagnosis to 60 days after MM diagnosis
  * early SREs if patients experienced it in the period included within 2 months after MM diagnosis up to 12 months
  * late SREs if patients experienced it in the period included within 12 months after MM diagnosis up to 24 months

SECONDARY OUTCOMES:
Number pf patients who suffered pain and its location | between 60 days before MM diagnosis and 60 days after MM diagnosis
  Pain will be collected evaluating clinical database, considering the situation at MM diagnosis
Number of patients with bone involvement at MM diagnosis | between 60 days before MM diagnosis and 60 days after MM diagnosis
  Describe any bone involvement including which bones. Data will be collected from clinical database, considering the situation at diagnosis.
Number of patients needing aids or orthoses | between 60 days before MM diagnosis and 24 months after MM diagnosis
  In the first 24 months after diagnosis, the use of aids or orthoses will be collected from clinical database. If possible the duration (in months) of use of aids or orthoses will be collected.
Number of patients who underwent therapy with zoledronic acid or other Bone Modifying Agents (BMAs) | between 60 days before MM diagnosis and 24 months after MM diagnosis
  The number of patients who received therapy with BMAs will be detected, considering the first 24 months from mm diagnosis.
Number of patients who received a Multiple Myeloma Multidisciplinary Team evaluation | period including 60 days before MM diagnosis and 24 months after diagnosis
  Data will be collected from clinical database, in the period including 60 days before MM diagnosis and 24 months after diagnosis. If a patient received more than 1 multidisciplinary team evaluation, this will be recorded
Number of patient who received a physiatric consultation | period including 60 days before MM diagnosis and 24 months after diagnosis
  Data will be collected from clinical database, in the period including 60 days before MM diagnosis and 24 months after diagnosis.
Number of patients who received a Rehabilitation intervention | period including 60 days before MM diagnosis and 24 months after diagnosis
  if the patient undergone to rehabilitation intervention, the study will describe:
  * Content of rehabilitation sessions
  * Number of sessions
  * Treatment goals
  * Any adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Fugazzaro, Physiatrist, Principal Investigator — AUSL-IRCCS of Reggio Emilia
Locations (1):
- AUSL-IRCCS of Reggio EmiliaOperational Unit of Physical Medicine and Rehabilitation AUSL - IRCCS Reggio Emilia, Reggio Emilia, Emilia Romagna 42123, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No